CLINICAL TRIAL: NCT03472573
Title: A Phase I Trial of Palbociclib in Combination With Dexamethasone in Relapsed or Refractory Adult B-Cell Acute Lymphoblastic Leukemia (ALL)
Brief Title: Palbociclib and Dexamethasone in Treating Participants With Relapsed or Refractory B-Cell Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17P.676; JT 11586 (Other: JeffTrial Number)
Record Dates: First submitted 2018-03-14; First posted 2018-03-21 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Recurrent B Acute Lymphoblastic Leukemia; Refractory B Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma | interventions — palbociclib; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (palbociclib, dexamethasone) (Experimental): INDUCTION: Participants receive palbociclib PO daily and dexamethasone PO daily for 28 days in the absence of disease progression or unacceptable toxicity. Participants with disease response (M0, M1, or M2) continue to Maintenance. Patients without a disease response discontinue treatment.
  MAINTENANCE: Participants receive dexamethasone with a taper PO daily on days 1-7. Participants also receive palbociclib daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Palbociclib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Palbociclib — Given PO
  Other Names: 571190-30-2; 6-Acetyl-8-cyclopentyl-5-methyl-2-((5-(piperazin-1-yl)pyridin-2-yl)amino)-8h-pyrido(2,3-d)pyrimidin-7-one; Ibrance; PD-0332991
Drug: Dexamethasone — Given PO
  Other Names: Baycuten; Cortidexason; Decacort; Desamethasone; Gammacorten; Loverine; Millicorten; Visumetazone

SUMMARY:
This phase I trial studies the side effects and best dose of palbociclib when given together with dexamethasone in treating participants with B-cell acute lymphoblastic leukemia that has come back after a period of improvement or does not respond to treatment. Palbociclib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Dexamethasone is a steroid medication that is used in combination with other medications to treat B-cell acute lymphoblastic leukemia. Giving palbociclib together with dexamethasone may work better in treating patients with B-cell acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the dose and schedule of the combination of palbociclib and dexamethasone in patients with relapsed or refractory adult B-cell acute lymphoblastic leukemia (ALL).

ii. To determine the safety and tolerability of the combination of palbociclib and dexamethasone in patients with relapsed or refractory adult B-cell ALL.

SECONDARY OBJECTIVES:

I. To evaluate the activity of palbociclib in combination with dexamethasone in patients with relapsed or refractory B-cell ALL.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologic evidence of relapsed or refractory B-cell ALL
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less
* Philadelphia chromosome positive (Ph+) patients must be refractory to or intolerant of standard tyrosine kinase inhibitor therapy
* Patients must be able to consume oral medication
* Patients must have recovered to =< grade 1 or stabilized from the toxic effects of any prior chemotherapy (except alopecia)
* Creatinine clearance (CrCL) >= 60 mL/min/1.73 m^2 calculated by Cockcroft-Gault
* Total bilirubin < 1.5 x upper limit of normal (ULN)
* Negative serum or urine pregnancy test for women with child-bearing potential
* Patients must be able to sign consent and be willing and able to comply with scheduled visits, treatment plan, procedures, and laboratory testing

Exclusion Criteria:

* Patients must not have evidence of active central nervous system (CNS) disease
* Patients must not be receiving any chemotherapy agents (except hydroxyurea); intrathecal methotrexate and intrathecal cytarabine are permissible
* Patients must not be receiving growth factors (granulocyte colony-stimulating factor [G-CSF], granulocyte-macrophage colony-stimulating factor [GM-CSF]), except for erythropoietin
* Patient must not have a concurrent active malignancy for which they are receiving treatment.
* Patients with other severe concurrent disease which in the judgment of the investigator would make the patient inappropriate for entry into this study are ineligible
* Patients must not have received any investigational agents within 30 days of study entry unless they have exceeded 5 terminal half-lives of the previous study drug used for treatment
* Patients must not be pregnant or breastfeeding; pregnancy tests must be obtained for all females of child-bearing potential within 10 days prior to enrollment; males or women of childbearing potential may not participate unless they have agreed to use an effective contraceptive method (defined as hormonal contraceptives, intrauterine devices, surgical contraceptives, or condoms)
* Patients who have uncontrolled infection are not eligible; patients must have any active infections under control; fungal disease must have been adequately treated for at least 2 weeks before study entry; subjects with bacteremia must have documented negative blood cultures prior to study entry
* Patients who are candidates for allogeneic transplantation, have a suitable donor, and are willing to undergo transplantation
* Patients who are eligible for and willing to receive treatment with tisagenlecleucel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2021-08-04 (Actual); Study Completion 2022-06-09 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLT) of the combination of palbociclib and dexamethasone | Up to 28 days after discontinuation of palbociclib and dexamethasone
  Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 should be used for grading.
Maximum tolerated dose (MTD) of the combination of palbociclib and dexamethasone defined as the highest dose level where a DLT occurs in at most one out of six patients treated | Up to 28 days after discontinuation of palbociclib and dexamethasone
  CTCAE version 4.03 should be used for grading.

SECONDARY OUTCOMES:
Clinically relevant responses to therapy determined by bone marrow biopsy | Up to 1 year
  Response rate defined as the proportion of patients who achieve an M, M1, or M2 response will be estimated along with a 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Kasner, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/73/NCT03472573/Prot_SAP_000.pdf